CLINICAL TRIAL: NCT01176539
Title: How Does the New Kai R Spot 100 Respiratory Monitor Compare to the Currently Used Respiratory Monitor for Measuring Respiratory Rate During Overnight Sleep Studies?
Brief Title: Substantial Equivalence Study for Kai Medical Non-Contact Respiratory Rate Monitor
Status: Completed | Type: Observational
Sponsor: Kai Medical, Inc. (Industry)
Responsible Party: Bob Nakata, Chief Technology Officer, Kai Medical, Inc.
Other Study IDs: KAI-00005; 18324 (Other: Stanford University)
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Respiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleep Clinic
  Interventions: Device: Non-Contact Respiratory Rate Monitor

INTERVENTIONS:
Device: Non-Contact Respiratory Rate Monitor — The Non-Contact Respiratory Rate Monitor provides a measurement of respiratory rate at a single point in time for neonates, pediatrics and adults.
  The Non-Contact Respiratory Rate Monitor provides a continuous monitor, measurement, and display of the respiratory rate, respiratory patterns, depth of breath, history/events and respiratory activity of a subject for neonates, pediatrics, and adults.

SUMMARY:
The purpose of this study is to determine whether the respiratory rate provided by Kai Medical Non-Contact Respiratory Rate Monitors are as accurate as that provided by the currently used methods, including respiratory chest bands.

ELIGIBILITY:
Inclusion Criteria:

* Every patient undergoing an overnight polysomnography study can be included.

Exclusion Criteria:

* None

Min Age: 29 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects at the Sleep Center at Stanford Universoty
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-03; Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Sleep Medicine Center, Redwood City, California, United States